CLINICAL TRIAL: NCT03714477
Title: A Prospective Randomized Study to Investigate the Effect of Extracorporeal Shockwave Lithotripsy on Blood Pressure Control in Patients With Hypertension - a Pilot Study
Brief Title: A Study to Investigate the Effect of Extracorporeal Shockwave Lithotripsy on Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Clinical Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRE 2018.276
Record Dates: First submitted 2018-10-15; First posted 2018-10-22 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Hypertension; Renal Stone
Keywords: Worsening hypertension; Renal stone
MeSH Terms: conditions — Hypertension; Nephrolithiasis | interventions — Lithotripsy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Active Comparator): immediate extracorporeal shock wave lithotripsy - subject will have SWL arranged in the next available list
  Interventions: Procedure: Extracorporeal shock wave lithotripsy
- Control Arm (No Intervention): delayed extracorporeal shock wave lithotripsy - subject will have SWL done 6 months later

INTERVENTIONS:
Procedure: Extracorporeal shock wave lithotripsy — A minimally invasive treatment for renal stone which was first introduced in early 1980's. It tries to fragment the renal stones by high-energy shockwave at the kidney from the outside.
  Arms: Treatment Arm

SUMMARY:
Having the advantages of being minimally invasive and simple, extracorporeal shock wave lithotripsy (SWL) remains one of the treatment options for renal stones less than 2cm. Although SWL is the most minimally invasive surgical approach for stone, there are still some concern about its short and long term side effect. While, there are some evidences that SWL might lead to increase in new onset hypertension, investigator's recent study suggested it might also cause worsening of blood pressure control in patient with known hypertension. Therefore, further studies are needed to confirm the initial finding. This study recruits patients who have hypertension and are currently diagnosed to have renal stone and planned for SWL, in order to to investigate the effect of SWL on blood pressure control.

After informed consent and background information have been obtained, patients will be randomized to either have routine SWL (treatment arm) or 6 months later (control arm). Group 1 patients will have blood pressure monitored for one day at home by an handy automated blood pressure measuring machine before SWL and 6 months after SWL. Group 2 patients will have blood pressure monitoring immediately and then 6 months later, just prior to the SWL.

DETAILED DESCRIPTION:
BACKGROUND

Extracorporeal shock wave lithotripsy (SWL) was first introduced in early 1980's for the management of urolithiasis. The advantage of being minimally invasive, when compared to other procedures for stone treatment, made SWL remain one of the treatment options for renal stones less than 2 cm in the latest guidelines.

Despite considered as the most non-invasive treatment for urinary calculi, there are still many concerns about the long-term consequence of SWL. In particular, the effect of SWL on blood pressure is still a controversy topic. In the recent study, investigator has observed approximately 20% of subjects experienced worsened blood pressure control during the 2-year follow-up period, including 20/202 (9.95%) previously non-hypertensive subjects who developed new onset hypertension. The observed incidence of new-onset hypertension was quite similar those in some reported series. In the literature, there were multiple reports, including case series and hospital data analyses, 7-9 of development of new-onset hypertension after SWL. Unfortunately, most of those studies were retrospective and used different definitions of hypertension.

But the high incidence of worsening blood pressure control, including 43 (36.4%) of 118 hypertensive subjects who required add-on antihypertensive therapies, observed in our study was alarming. Because most studies in the literature were just focused on development of new-onset hypertension, investigator's observation provides supplementary information about potential effects of SWL on pre-existing hypertension. In general, the average annual incidence of add-on pharmacotherapy among local hypertensive patients was 4.71-6.41%. 10 Therefore, the add-on therapy rate of 36.4% during the 2-year follow-up was much higher than that in the general population. Unfortunately, investigator did not include a non-interventional arm for comparison in the previous study and could not conclude that this outcome was solely attributable to SWL.

Therefore, investigator would like to propose a prospective study to assess the effect SWL on the blood pressure control in patients with known hypertension. Investigator hope the study results will provide additional information on the long-term effect of SWL on patients.

OJECTIVES

To investigate the effect of extracorporeal shockwave lithotripsy on the effect of change in blood pressure in patients with known hypertension.

STUDY PROTOCOL:

Patients fulfilled the inclusion and exclusion criteria specific to this study will be prospectively recruited. After obtaining informed consent, patients will be randomized to either treatment group or control group.

Baseline information, including age, years of diagnosed to have hypertension, current medical usage, other comorbidities, BMI etc. will be collected from patients. All SWL would be performed in the Lithotripsy and Uro-investigation Centre of the Prince of Wales Hospital, and treated by Modulith SLX-F2 Connect (Storz Medical, Switzerland), an electromagnetic lithotriptor. The treatment would be performed as standard care in our hospital. After SWL, the patient would be follow-up in clinic as usual. During the 6 months study period, patients are strongly advised to avoid change in hypertensive medication.

Blood pressure assessment:

During each blood pressure assessment, the following procedure will be performed:

1. 24-hour blood pressure monitoring - 24-h non-invasive ambulatory BP and HR monitoring was performed using a validated device and followed the recommended approached. 11 The blood pressure measurement would be programmed to measure BP every 15 min. Each recording will be started in the morning and performed throughout a full 24-h period, during which subjects are allowed to follow their normal daily routine. The analysis of 24-h BP recordings are preceded by removal of artifacts, according to previously described editing criteria. 12 Recordings are excluded from the analysis when > 10% of all readings or more than one reading per hour is missed. Computed analysis of the individual recordings provided 24-h, night-time (23.00-07.00 h), morning-time (0.7.00-12.00 h), and afternoon/evening-time (12.00- 23.00 h) mean values of SBP, DBP, and HR.
2. Clinic blood pressure measurement At each visit, blood pressure will be measured after patient rested for more than 10 minutes, with repeated measurement 5 minutes apart. The mean blood pressure will be recorded.
3. Any changes in antihypertensive drugs and reasons
4. Any adverse events.

The result collected will be used for further analysis

ELIGIBILITY:
Inclusion Criteria:

* Renal calculi of size 5-15 mm in maximal diameter and considered as suitable for SWL
* Patient with known hypertension and on regular medical treatment with regular follow-up.
* Patient with stable hypertension for at least 3 months

Exclusion Criteria:

* Patients had previous SWL, kidney surgery, percutaneous nephrolithotomy, etc.
* Patients with stones obviously required more than one section of SWL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
The changes in mean 24hr systolic and diastolic blood pressure measurement | Baseline, 6 months
  For treatment arm, the changes in mean 24hr systolic and diastolic blood pressure measurement before SWL and 6 monthes after SWL For control arm, the changes in mean 24hr systolic and diastolic blood pressure measurement right after randomization and in 6 months.

SECONDARY OUTCOMES:
Change in mean night time diastolic and systolic blood pressure | Baseline, 6 months
  For treatment arm, the changes in mean night time systolic and diastolic blood pressure measurement before SWL and 6 monthes after SWL For control arm, the changes in mean night time systolic and diastolic blood pressure measurement right after randomization and in 6 months.
Change in mean night time heart rate | Baseline, 6 months
  For treatment arm, the changes in mean heart rate before SWL and 6 monthes after SWL For control arm, the changes in mean night time heart rate right after randomization and in 6 months.
Change in mean morning-time diastolic and systolic blood pressure | Baseline, 6 months
  For treatment arm, the changes in mean morning-time systolic and diastolic blood pressure measurement before SWL and 6 monthes after SWL For control arm, the changes in mean morning-time systolic and diastolic blood pressure measurement right after randomization and in 6 months.
Change in mean morning-time heart rate | Baseline, 6 months
  For treatment arm, the changes in mean morning-time heart rate before SWL and 6 monthes after SWL For control arm, the changes in mean morning-time heart rate right after randomization and in 6 months.
Change in mean afternoon/evening diastolic and systolic blood pressure | Baseline, 6 months
  For treatment arm, the changes in mean afternoon/evening systolic and diastolic blood pressure measurement before SWL and 6 monthes after SWL For control arm, the changes in mean afternoon/evening systolic and diastolic blood pressure measurement right after randomization and in 6 months.
Change in mean afternoon/evening heart rate | Baseline, 6 months
  For treatment arm, the changes in mean afternoon/evening heart rate before SWL and 6 monthes after SWL For control arm, the changes in mean afternoon/evening heart rate right after randomization and in 6 months.
Change in mean 24hr heart rate | Baseline, 6 months
  For treatment arm, the changes in mean 24hr heart rate measurement before SWL and 6 monthes after SWL For control arm, the changes in mean 24hr heart rate measurement right after randomization and in 6 months.
The need of add-on therapy for hypertension | 6 months
  Any add-on anti-hypertensive drugs in 6 months time
Any adverse effects after SWL | 6 months
  Any adverse effects comparing the treatment arm and control arm during study period

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, Md, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
No individual participant data will be shared to other researchers outside CUHK Urology unit